CLINICAL TRIAL: NCT00916331
Title: Subcutaneous Indwelling of Vacuum Drainage in Total Knee Arthroplasty: Prospective Randomized Comparisons With Intraarticular Indwelling
Brief Title: Subcutaneous Indwelling of Vacuum Drainage in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Tae Kyun Kim, Joint Recontruction Center, Seoul National University Bundang hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-0606/034-008
Record Dates: First submitted 2009-05-15; First posted 2009-06-09 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Total Knee Arthroplasty
Keywords: total knee replacement arthroplasty; subcutaneous indwelling; blood loss; complications; functional status
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- subcutaneous group (Experimental): Vacuum drainage is indwelled in subcutaneous layer
  Interventions: Procedure: subcutaneous indwelling
- intraarticular group (Experimental): Vacuum drainage is indwelled in intraarticular space
  Interventions: Procedure: intraarticular indwelling

INTERVENTIONS:
Procedure: subcutaneous indwelling — vacuum drainage is indwelled in subcutaneous layer
  Other Names: hemovac
  Arms: subcutaneous group
Procedure: intraarticular indwelling — vacuum drainage is indwelled in intraarticular space
  Other Names: hemovac
  Arms: intraarticular group

SUMMARY:
This prospective, randomized trial asked whether subcutaneous indwelling of vacuum drainage has advantages over intraarticular indwelling in terms of blood loss, bleeding related complications, and functional outcomes in primary total knee arthroplasty (TKA). The investigators hypothesized that the subcutaneous indwelling method would reduce blood loss with comparable bleeding-related complications and functional outcomes. The subcutaneous indwelling group demonstrated reduced blood loss with comparable prevalence of bleeding-related complications and functional outcomes. In conclusion, the investigators' study verified the efficacy and absence of risks of subcutaneous indwelling method. So the investigators propose that the subcutaneous indwelling drainage can be a good option to address the problems related to postoperative bleeding after TKA.

DETAILED DESCRIPTION:
There are numerous reports in the literature on drainage options after TKA, but there is no consensus. Many studies have shown no apparent advantage of drainage but routine intraarticular indwelling drainage after TKA has been extensively used to avoid complications associated with hematoma formation. It is of interest to determine if it is possible to reduce blood loss while still using drainage. So we came to think about a new and more convenient method-subcutaneous indwelling. Theoretically subcutaneous indwelling method which still has the advantages over the intraarticular indwelling method but is more convenient than drain-clamping method may be a better option. So we hypothesized that subcutaneous indwelling method of vacuum drainage has advantages over the intraarticular indwelling method.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis
* primary total knee arthroplasty
* Signed written informed consent
* Spinal/epidural anesthesia

Exclusion Criteria:

* Patients with coagulation disorders
* Revision total knee arthroplasty
* Simultaneous bilateral total knee arthroplasty
* Diagnosis other than primary osteoarthritis
* Patients refusing consents

Ages: 54 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
blood parameters by which we can estimate blood loss , such as drained blood volume, hemoglobin and hemoglobin drop | 24 hours after operation

SECONDARY OUTCOMES:
transfusion | during hospital stay
wound problem | during hospital stay
hypotension episode | during hospital stay
functional outcome (ROM, AKS Knee score, WOMAC score, SF-36 score) | preoperative & postoperative 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyun Kim, MD, PhD, Principal Investigator — Joint Recontruction Center, Seoul National University Bundang hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea